CLINICAL TRIAL: NCT00400010
Title: Randomized Controlled Trial of a Expert System for Patients With At-risk Drinking, Alcohol Abuse and Alcohol Dependence in General Hospital
Brief Title: Alcohol Expert System Intervention for Problematic Alcohol Use
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Luebeck (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government)
Responsible Party: Principal Investigator, Hans-Jürgen Rumpf, PD Dr. Hans-Jürgen Rumpf, University of Luebeck
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 01EB0421-1
Record Dates: First submitted 2006-11-14; First posted 2006-11-16 (Estimated); Last update posted 2014-04-02 (Estimated); Status verified 2014-04

CONDITIONS: Alcohol-related Disorders; Alcohol Drinking
Keywords: Expert system; Transtheoretical Model of Behavior Change; Brief intervention; General hospital
MeSH Terms: conditions — Alcohol-Related Disorders; Alcohol Drinking

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Expert System Intervention (Experimental): Computerized Expert System Intervention based on the Transtheoretical Model of Change: 1. Normative feedback and feedback on motivational variables during the first week of hospital stay 2. Ipsative feedback on drinking behavior and motivation to change after three months
  Interventions: Behavioral: Expert System Intervention
- Control group (No Intervention): Controls received a brochure on health behavior

INTERVENTIONS:
Behavioral: Expert System Intervention — Questionnaires on motivation to change and alcohol consumption were assessed in a clinical interview. Data were entered in a Computer and a fully automatized feedback letter was generated by an expert system. The printed feedback letter was handed out to patients by study staff the following day.
  Arms: Expert System Intervention

SUMMARY:
In a randomized controlled trial, patients recruited in a general hospital and fulfilling criteria for alcohol dependence, alcohol abuse or at-risk drinking will be randomly allocated to two conditions:(1) Transtheoretical Model (TTM)-based expert system group, patients receive an individualized feedback on drinking norms, health-related risks and core constructs of the TTM, augmented by a TTM-based manual, (2) Control group,receiving a booklet on health behavior.

Outcome assessment will be conducted after 12 months. The hypothesis is that individualized feedback leads to greater reduction in alcohol consumption and elevated readiness to change at follow-up.

DETAILED DESCRIPTION:
Background: A promising approach in secondary prevention of problem drinking is to provide brief interventions in medical settings. However, brief interventions have not become implemented in general practices (GPs) due to insufficient role security and therapeutic commitment of physicians. Computerized expert systems can provide very cost-effective means of intervention and have been effective in the field of smoking cessation. However, in the alcohol field, research on this issue is scarce.

Objectives: Comparing an expert system based on the Transtheoretical Model of behavior change for patients with at-risk drinking, alcohol abuse or alcohol dependence to a control condition. Methods: About 2,500 screenings among consecutive general hospital patients aged 18 to 64 will be conducted. Subjects fulfilling inclusion criteria (severe alcohol dependence excluded) will be randomly assigned to one of two conditions with 150 patients each: (1) In the TTM-based expert system group, patients receive an individualized feedback on drinking norms, health-related risks and core constructs of the TTM, augmented by a TTM-based manual. (2) In the control group, participants receive a booklet on health behavior. Outcome assessment will be conducted after 12 months. Outcome variables are alcohol consumption, stages of change progress and utilization of formal help. Expected impact: Findings are expected to provide evidence for a computerized TTM based expert system to be used in primary care. This would be the first international results confirming such an approach in the alcohol field. If a TTM-based expert system would be effective, this could significantly save resources and enhance secondary prevention. Therefore, data are of great public health interest. Relationship to the objective of the collaboration: As in the other studies, empirical data on new proactive approaches to reach underserved populations in the addiction field will be provided. The project will add knowledge on the economical use of interventions.

ELIGIBILITY:
Inclusion Criteria:

* Alcohol Abuse
* Alcohol Dependence
* At-risk drinking

Exclusion Criteria:

* Current treatment for alcohol problems
* Terminal illness

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 347 (Actual)
Dates: Start 2004-10; Primary Completion 2005-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Average alcohol consumption (QF) gr/alc. per day | 12 months
  Main outcome is reduction in daily average alcohol consumption, operationalized by a Quantity-/Frequency measure

SECONDARY OUTCOMES:
Readiness to change drinking behavior | 12 months
  Readiness to change questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Hans-Juergen Rumpf, Ph.D., Principal Investigator — University of Luebeck
Locations (1):
- University of Luebeck, Dpt. of Psychiatry and Psychotherapy, Lübeck, Germany

REFERENCES:
- [Derived] Bischof G, Freyer-Adam J, Meyer C, John U, Rumpf HJ. Changes in drinking behavior among control group participants in early intervention studies targeting unhealthy alcohol use recruited in general hospitals and general practices. Drug Alcohol Depend. 2012 Sep 1;125(1-2):81-8. doi: 10.1016/j.drugalcdep.2012.03.018. Epub 2012 Apr 18. PMID 22516146